CLINICAL TRIAL: NCT01498978
Title: A Phase II Study of CTLA Blockade by Ipilimumab Plus Androgen Suppression Therapy in Patients With an Incomplete Response to AST Alone for Metastatic Prostate Cancer
Brief Title: Ipilimumab in Combination With Androgen Suppression Therapy in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Julie Graff, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00005254; NCI-2011-03556 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CA184059 (Other Grant/Funding Number: Bristol-Myers Squibb Company Protocol Number); 08-004 (Other: Prostate Cancer Clinical Trials Consortium Protocol Number); 5254 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ipilimumab) (Experimental): Patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients without progression then receive maintenance ipilimumab IV once every 3 months for 4 additional doses.
  Interventions: Biological: ipilimumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: ipilimumab — Given IV
  Other Names: anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody; MDX-010; MDX-CTLA-4; monoclonal antibody CTLA-4
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well ipilimumab works when given together with androgen suppression therapy in treating patients with hormone-resistant prostate cancer that has spread to other parts of the body. Monoclonal antibodies, such as ipilimumab, can block tumor growth in different ways. Some block the ability of tumors to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Androgen can cause the growth of prostate cancer. Androgen deprivation therapy may stop the adrenal glands from making androgen. Giving ipilimumab together with androgen suppression therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Proportion of patients who achieve an undetectable prostate-specific antigen (PSA) (=< 0.2 ng/ml) after initiation of ipilimumab therapy.

SECONDARY OBJECTIVES:

I. Time to PSA progression. II. Time to progression by any measure. III. Maximum percentage of PSA reduction in each patient. IV. Number of patients with immune related adverse events (IRAEs) and correlation of these with complete PSA response, time to progression, and T cell measurements.

V. Measures of T cell response to therapy with flow cytometry. VI. Response in measurable disease by modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

VII. Time to death from any cause. VIII. To examine correlative biomarkers and their relationship to clinical outcomes. Potential biomarkers include, but are not limited to C-reactive protein (CRP), insulin-like growth factor (IGF)-1 and -2, or follicle stimulating hormone (FSH).

XV. Bank samples for future molecular correlative studies, biomarker, or other studies.

OUTLINE:

Patients receive ipilimumab intravenously (IV) over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients without progression then receive maintenance ipilimumab IV once every 3 months for 4 additional doses.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Histologic diagnosis of adenocarcinoma of the prostate
* A PSA of > 0.2 ng/ml after 6-18 months of androgen suppression therapy, which may consist of luteinizing hormone-releasing hormone (LHRH) agonist or antagonist alone or the combination of an LHRH agonist or antagonist plus an antiandrogen, such as bicalutamide; androgen suppression therapy will continue without interruption
* Radiographic evidence of regional or distant metastasis at the time of study enrollment or at the time of diagnosis
* White blood cell (WBC) >= 2000/uL
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets >= 50 x 10^3/uL
* Hemoglobin >= 8 g/dL
* Creatinine =< 3.0 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN for patients without liver metastasis
* Bilirubin =< 3.0 x ULN, (except patients with Gilbert's syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* No known active or chronic infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; patients should be assessed for high risk behaviors that may result in these infections, such as intravenous drug use or multiple sexual partners; the assessment should be noted
* Eastern Cooperative Oncology Group (ECOG) =< 1
* Patients receiving any herbal product known to decrease PSA levels (i.e. saw palmetto and prostate cancer [PC]-SPES), or any immunosuppressive dose of systemic or absorbable topical corticosteroid (except prednisone up to 10 mg orally per [q] day, or its equivalent), must discontinue the agent for at least 2 weeks prior to screening; progressive disease must be documented after discontinuation of these products
* Patients receiving bisphosphonate therapy must have been on stable doses for at least 4 weeks with stable symptoms prior to the first infusion with ipilimumab
* Total testosterone < 50 ng/ml, except in patients with prior orchiectomy, where testosterone does not need to be measured; patients must continue their LHRH agonist therapy throughout study duration
* Life expectancy >= 6 months; this must be documented
* Patients who are sexually active with a partner who could become pregnant are to use an effective form of barrier contraception, such as condoms or a partner using oral contraceptive pills; persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 8 weeks after ipilimumab is stopped
* If a patient enters the trial on androgen suppression therapy (AST) that consists of both an LHRH agonist and an oral antiandrogen, both agents should be continued throughout the study; if an antiandrogen is stopped prior to study entry, it should be stopped 4 weeks before for nilutamide and flutamide and 6 weeks before for bicalutamide to ensure that a withdrawal phenomenon does not interfere with interpretation of efficacy results

Exclusion Criteria:

* Radiation to any area of the body < 28 days prior to randomization
* Any other active malignancy with the exception of adequately treated basal or squamous cell skin cancer or superficial bladder cancer
* Autoimmune disease: patients with a history of inflammatory bowel disease are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. myasthenia gravis, Guillain-Barre syndrome); those with immune-mediated skin toxicity (i.e. toxic epidermal necrolysis, Stevens-Johnson syndrome) will also be excluded
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab)
* A history of prior treatment with ipilimumab or prior cluster of differentiation (CD)137 agonist or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitor or agonist
* Concomitant therapy with any of the following: interleukin (IL)-2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents (over the counter [OTC]/herbal/prescribed); immunostimulant agents, other than the study agent; other investigational therapies; or chronic use of systemic corticosteroids (greater than prednisone 10 mg orally per day, or its equivalent)
* Prisoners or patients who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (i.e., infectious) illness

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02-06 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2019-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Graff, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - OHSU Knight Cancer Institute, Portland, Oregon

REFERENCES:
- [Derived] Graff JN, Stein MN, Surana R, Al Rabadi L, Liu E, Fong L, Bailey S, Latour E, Newby TA, Moran AE, Beer TM. Phase II Study of Ipilimumab in Men With Metastatic Prostate Cancer With an Incomplete Response to Androgen Deprivation Therapy. Front Oncol. 2020 Aug 7;10:1381. doi: 10.3389/fonc.2020.01381. eCollection 2020. PMID 32850444

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ipilimumab)
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: 10 subjects received combination therapy.
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 64.5 [56 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Achieve an Undetectable PSA (=< 0.2 ng/ml)
Description: Undetectable PSA (prostate-specific antigen) defined as PSA ≤ 0.2 ng/mg after initiation of ipilimumab therapy.
  Provided with the exact 95% confidence interval. PSA response as recommended by the Prostate Cancer Clinical Trials Working Group (PCWG2) definitions.
  Percentage can take on values between 0% and 100%.
Time Frame: Up to 5 years
Population: Intention to Treat (ITT) population -- all patients who sign the consent and are assigned to a treatment regardless of the actual drug dose the patients receive
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 10
percentage of patients | 0.0 [0.0 to 0.0]

2. Secondary Outcome: Time to PSA Progression
Description: PSA (prostate-specific antigen) progression defined as a PSA increase of >= 25% and at least 2 ng/mL from baseline or nadir PSA achieved, confirmed by a second measurement at least three weeks later
  Time to PSA progression is calculated as the time from Day 1 of combination therapy to first PSA measurement of >= 25% increase and at least 2 ng/mL above the nadir and confirmed by a second measurement at least three weeks later. For subjects without a PSA decline from baseline, time to PSA progression is calculated as the time from Day 1 of combination therapy to first PSA measurement of >= 25% increase and at least 2 ng/mL increase from baseline after 12 weeks and confirmed by a second measurement at least three weeks later.
  Outcome is reported as median time to event determined by the Kaplan Meier method with 95% confidence interval.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 10
days | 525 [77 to NA] — Upper limit not able to be estimated.

3. Secondary Outcome: Time to Progression by Any Measure
Description: Time to progression is calculated from Day 1 of combination therapy to first evidence of progression by any measure (PSA, Measurable Disease or Clinical Progression).
  Outcome is reported as median time to event determined by the Kaplan Meier method with 95% confidence interval.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 10
days | 118 [63 to 532]

4. Secondary Outcome: Time to Death From Any Cause
Description: Time to death is calculated from Day 1 of combination therapy to death from any cause.
  Outcome is reported as median time to event determined by the Kaplan Meier method with 95% confidence interval.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 10
days | 1825 [470 to NA] — Upper limit not able to be estimated.

5. Secondary Outcome: Number of Patients With IRAEs
Description: Immune-Related Adverse Events (IRAEs) are defined as an adverse event (AE) of unknown etiology associated with drug exposure and consistent with an immune phenomenon
  Tabulated for each treatment group and summarized according to major organ categories of the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ipilimumab)
Number analyzed (Participants) | 10
Participants | 6
Statistical Analysis 1: Comparison: Treatment (Ipilimumab); Exact binomial test (two-sided). Null hypothesis: the proportion is equal to 0.5; Test type: Other — Exact binomial test (two-sided); p = 0.754, Exact Binomial Test

6. Secondary Outcome: Correlation Between IRAE and PSA Progression.
Description: Immune related adverse event (IRAE) is defined as any adverse event associated with drug exposure and consistent with an immune-mediated event. PSA (prostate-specific antigen) Progression is defined as a PSA increase of >= 25% and at least 2 ng/mL from Baseline, or Nadir PSA Achieved, confirmed by a second measurement at least three weeks later.
  The correlation between IRAEs and clinical outcomes will be evaluated using logistic regression for binary endpoints and Cox regression for the time to event outcomes. Due to sample size, regression is not feasible. Instead, correlation will be assessed by Fishers Exact test of association.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Yes: IRAE: Patients that experienced an IRAE.
  Immune related adverse event (IRAE) is defined as any adverse event associated with drug exposure and consistent with an immune-mediated event.
- No: IRAE: Patients that did not experience an IRAE.
  Immune related adverse event (IRAE) is defined as any adverse event associated with drug exposure and consistent with an immune-mediated event.
Arm/Group | Yes: IRAE | No: IRAE
Number analyzed (Participants) | 6 | 4
Participants
  Yes: PSA Progression | 5 | 1
  No: PSA progression | 1 | 3
Statistical Analysis 1: Comparison: Yes: IRAE vs No: IRAE; Test type: Other — Test of association (contingency) between the two kinds of classification; p = 0.190, Fisher Exact

7. Secondary Outcome: Correlation of IRAEs With Ratio of T Regulatory Cells to T Effector Cells
Description: Immune related adverse event (IRAE) is defined as any adverse event associated with drug exposure and consistent with an immune-mediated event.
  Raw T cells data was collected, but has not been analyzed by the lab and will not be done due to constraints.
  No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Up to day 1 of course 4
Population: as for outcome 1
Arm/Group | Yes: IRAE | No: IRAE
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Correlation Between IRAEs and Immune Response
Description: Immune related adverse event (IRAE) is defined as any adverse event associated with drug exposure and consistent with an immune-mediated event.
  Outcome not evaluated due to technical challenges collecting the data, and lack of budget and personnel to complete the analysis.
  No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Up to day 1 of course 4
Population: as for outcome 1
Arm/Group | Yes: IRAE | No: IRAE
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Correlation Between IRAE and Radiographic Progression.
Description: Immune related adverse event (IRAE) is defined as any adverse event associated with drug exposure and consistent with an immune-mediated event. Radiographic progression is progression determined by scan.
  The correlation between IRAEs and clinical outcomes will be evaluated using logistic regression for binary endpoints and Cox regression for the time to event outcomes. Due to sample size, regression is not feasible. Instead, correlation will be assessed by Fishers Exact test of association.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Yes: IRAE | No: IRAE
Number analyzed (Participants) | 6 | 4
Participants
  Yes: Radiographic progression | 1 | 2
  No: Radiographic progression | 5 | 2
Statistical Analysis 1: Comparison: Yes: IRAE vs No: IRAE; Test type: Other — Test of association (contingency) between the two kinds of classification; p = 0.500, Fisher Exact

10. Secondary Outcome: Correlation Between IRAE and Any Progression.
Description: Immune related adverse event (IRAE) is defined as any adverse event associated with drug exposure and consistent with an immune-mediated event.
  The correlation between IRAEs and clinical outcomes will be evaluated using logistic regression for binary endpoints and Cox regression for the time to event outcomes. Due to sample size, regression is not feasible. Instead, correlation will be assessed by Fishers Exact test of association.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Yes: IRAE | No: IRAE
Number analyzed (Participants) | 6 | 4
Participants
  Yes: Any progression | 5 | 3
  No: Any progression | 1 | 1
Statistical Analysis 1: Comparison: Yes: IRAE vs No: IRAE; Test type: Other — Test of association (contingency) between the two kinds of classification; p = 1.000, Fisher Exact

11. Secondary Outcome: Correlation Between IRAE and Overall Survival.
Description: as for outcome 10
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Yes: IRAE | No: IRAE
Number analyzed (Participants) | 6 | 4
Participants
  Yes: Deceased | 2 | 3
  No:Deceased | 4 | 1
Statistical Analysis 1: Comparison: Yes: IRAE vs No: IRAE; Test type: Other — Test of association (contingency) between the two kinds of classification; p = 0.524, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the start of Ipilimumab therapy until off study for progression, adverse event or other reason, an average of one year.
Description: Only Adverse Events that are considered possibly related or related to the study procedures or study drug are reported.
Arm/Group | Treatment (Ipilimumab)
All-Cause Mortality (participants affected / at risk) | 2/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ipilimumab) (N=10)
Diarrhea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ipilimumab) (N=10)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 6 (11)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 (4) — rash
Fatigue (General disorders) | 4 (4)
Fever (General disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Aspartate aminotransferase (Investigations) | 1 (2)
Alanine aminotransferase (Investigations) | 1 (2)
Alkaline phosphatase (Investigations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Dupuytren's Contracture
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT01498978/Prot_SAP_000.pdf